CLINICAL TRIAL: NCT05482373
Title: Nutraceuticals and Functional Foods of the Olive Tree of Interest in Aging and Its Pathologies: Study of Mechanisms of Action and Clinical Trial in Patients With Periodontitis
Brief Title: Adjuvant Treatment in Elderly Patients With Periodontitis Through the Administration of a Supplement Rich in Oleuropein From the Olive Leaf
Acronym: OLIVAGING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jose Luis Quiles Morales (Other)
Responsible Party: Sponsor-Investigator, Jose Luis Quiles Morales, Full Professor, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI-001-2020
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Periodontitis
Keywords: Aging; Periodontitis; Nutraceuticals; Oleuropein; Olive tree; Adjuvant
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive hard gelatin capsules containing placebo (only the excipients).
  Interventions: Dietary Supplement: Placebo
- Oleuropein (Experimental): Patients will receive the same hard gelatin capsules but containing 200 mg of an olive leaf extract.
  Interventions: Dietary Supplement: Oleuropein from olive tree

INTERVENTIONS:
Dietary Supplement: Oleuropein from olive tree — The capsules intake will last for a total of 4 months.
  Arms: Oleuropein
Dietary Supplement: Placebo — The capsules intake will last for a total of 4 months.
  Arms: Placebo

SUMMARY:
Life expectancy has dramatically increased in the last century, although this process has not been always accompanied by an equivalent increase in healthy life expectancy. However, extending longevity without decreasing the risk of age-associated pathologies would not be desirable since non-communicable diseases can diminish seniors' quality of life, raise health-care costs, and increase pressure on family members who are responsible for their care. Maintaining a good health would help to ensure independence, security, and continued productivity in the later years helping both health systems and pensions lower costs. Thus, many scientific studies have tried to delay the age of onset of major age-related chronic diseases. In other words, research has been more focused on extending healthspan rather than lifespan.

Actually, numerous experimental studies have shown that the extension of lifespan by modifying risk factors is usually accompanied by delayed or reduced morbidity, including cardiovascular disease, neurodegeneration, and tumors. In the dietary context, modifications of the diet energy and/or macronutrient balance has shown to contribute to healthy aging, increasing healthspan and probably lifespan. Likewise, some foods would be able to supply a significant amount of compounds to the human diet, including non-nutrients which are thought to exert effects in the same sense. Thus, adequate nutritional intervention would be considered geroprotective interventions that would positively influence health by slowing basic biological processes of aging, such as cellular senescence, mitochondrial dysfunction, age-related decline of stress resistance, dysregulated cellular energy sensing/growth pathways, impaired proteostasis, deteriorated stem cell function/bioavailability, as well as inflammation/oxidative stress.

The use of nutraceuticals and functional foods from olive products and by-products can be useful in the treatment of pathologies associated with aging, such as periodontitis, as well as from the point of view of a proper nutrition during aging.

The study is a double-blind clinical trial of parallel design whose main objective is to evaluate the usefulness of a dietary supplement rich in oleuropein from the olive tree (leaf) in the adjuvant treatment of patients with age-related periodontitis. Efforts will be made to ensure that men and women be represented homogeneously in all study groups, although it is known that gender does not influence the appearance of periodontitis.

The experimental design foresees the inclusion of 130 patients with chronic periodontitis aged 60 years or older, 65 for the control group and 65 for the treatment group. Volunteers will be recruited from new patients attending the Faculty of Odontology at the University of Sevilla, Sevilla (Spain) by one study team member.

The investigational product will be provided by Natac Company (Madrid, Spain), a corporate group dedicated to researching, developing, manufacturing, and marketing natural ingredients to be used in food supplements, feed, pet food, as well as in functional foods, and as natural, active pharmaceutical ingredients.

The planned schedule for the participating subjects is as follows:

* Day 0: diagnosis of periodontitis, proposal to participate in the study, delivery of consent and information to the patient.
* Day 15: oral exams, collection of sociodemographic data, study of anthropometric characteristics and blood pressure, evaluation of eating habits, urine and blood sampling, collection of samples for the study of the periodontal microbiota and data collection and calculation of the index of successful ageing.
* Day 16 to 30 periodontal treatment.
* Day 16 to 136: administration of treatment (oleuropein or placebo).
* Day 136: oral exams, collection of sociodemographic data, study of anthropometric characteristics and blood pressure, evaluation of eating habits, urine and blood sampling, collection of samples for the study of the periodontal microbiota and data collection and calculation of the index of successful ageing.

The analytical part of the of the clinical trial will be developed mostly in the Biomedical Research Center (CIBM) of the University of Granada. The field part of the clinical trial in patients with periodontitis will be carried out at the Faculty of Dentistry of the University of Seville.

The design of the clinical trial provides for the participation of specialists from several disciplines, including specialists in Nutrition and Physiology, clinical specialists in Pathological Anatomy and Dentistry, technicians from the Center of Scientific Instrumentation of the University of Granada (specialists in various subjects such as microscopy, biochemical analysis, histology and veterinary) as well as technicians from the Marketing Unit of the OTRI of the University of Granada.

DETAILED DESCRIPTION:
To calculate the sample size, the GRANMO tool (https://www.imim.es/ofertadeserveis/software-public/granmo/) has been used, considering an alpha risk of 0.05, a bilateral contrast, a beta risk of 0.20, a standard deviation of differences of 2.5, a minimum difference of 1 mm reduction in probing depth to be detected between baseline and end of study, and a predicted proportion of loss of 20% tracking.

Treatments All patients will receive a complete oral examination at baseline and after 4 months following the treatment. Initial therapy will be performed in all patients and will consist on full-mouth scaling and root planning by hand and with ultrasonic instrumentation as necessary. This treatment will be completed with oral hygiene instructions. All initial therapy procedures will be performed by the same periodontist.

After periodontal treatment, enrolled volunteers will be randomly assigned to one of two groups by a second periodontist. Control group will receive hard gelatin capsules containing placebo (only the excipients), whereas the experimental group will receive the same hard gelatin capsules but containing 200 mg of an olive leaf extract. The randomization will be done by the use of random number charts (by coin-toss), which will be performed at the time of the first subject's enrollment, and the next subject will be assigned to the other group based on the first subject's assignment. Both placebo and capsules will be dispensed by the same person, and subjects will be given verbal and written instructions on its use. As volunteers will be enrolled they will be allocated sequential study numbers and provided with their capsules, sufficient for one month. Subjects will come to the Faculty every 4 weeks during the course of the trial to replenish their capsules. The capsules intake will last for a total of 4 months. Remaining medications will be checked for compliance. Capsules will be prepared at the CIDAF (Centro de Investigación Sobre Alimentos Funcionales) at the Technological Health Park in Granada. The olive extract will be obtained from Natac company (Madrid, España).

Sample collection and analyses All data collection and determinations will be performed at baseline and after 4 months.

A) Oral examinations Periodontal clinical measurements will include the presence or absence of supragingival dental plaque and gingival bleeding on probing (BOP), as well as periodontal probing depth (PPD) and recession of the gingival margin (GM). Parameters will be measured at six sites (mesiobuccal, buccal, distobuccal, distolingual, lingual, and mesiolingual) on every tooth by means of a calibrated periodontal probe (Hu-Friedy®, Chicago, IL, USA), 15 mm in length and 0.35 mm in diameter. Clinical attachment level (CAL) will be calculated by adding recession to PDD. The number of remaining teeth will also be recorded. O´Leary's plaque index, Van der Velden's bleeding index will be also calculated. Patients with BOP site <10%, PPD ≤3 mm, erythema and edema absence will be considered periodontal-healthy subjects.

B) Sociodemographic data collection

1. Basic sociodemographic data: these will include age, gender, years of education.
2. Financial status: participants will be asked to report their mean income during the previous three years using a four-point scale (low, inadequate to cover daily expenses = 1, medium, trying hard to cover daily expenses = 2, good, adequate to cover daily expenses = 3, very good, very adequate to cover daily expenses = 4).
3. Smoking status: current smokers will be defined as smokers at the time of the interview. Former smokers will be defined as those who had previously smoked, but had not done so for a year or more. The remaining participants will be defined as occasional or non-current smokers.
4. Physical activity level: it will be evaluated in metabolic equivalent (MET)-minutes per week, using the self-reported International Physical Activity Questionnaire (IPAQ). Those who reported at least 3 MET-minutes per week will be classified as physically active (minimally active - or "health enhancing physical activity (HEPA) active"). All others will be defined as physically inactive. Furthermore, the weekly frequency of physical activity will be recorded.
5. Last month's depression symptoms: they will be assessed using a validated shortened, self-report Geriatric Depression Scale (GDS) (range 0-20). A GDS score between 0 and 4 will be used to indicate no depression, while scores of 5-10 and N 10, will indicate mild and severe depression, respectively.
6. Healthcare use: the presence of private physicians' offices, public or private health care centers or hospitals in the area of residence, as well as the annual number of visits for regular check-up of the health status, will be recorded.
7. Adult's social participation: weekly frequency of their social activities with their family, their friends as well as their yearly frequency of excursions will be recorded for this purpose.

C) Anthropometric characteristics and blood pressure

1. Weight, height and waist circumference will be measured. BMI and waist-to-hip ratio will be calculated. Overweight will be defined as BMI between 25.0 and 29.9 kg/m2, while obesity will be defined as BMI >29.9 kg/m2.
2. Blood pressure: patients with blood pressure levels>140/90 mmHg or using antihypertensive medications will be classified as hypertensive.

D) Dietary habits assessment The evaluation of dietary habits will be based on a semi-quantitative food-frequency questionnaire (FFQ). FFQ will be used to evaluate the level of adherence to the Mediterranean diet, the MedDietScore (theoretical range 0-55) was used.

E) Blood sampling and analysis Blood samples (16 mL) will be collected by forearm venipuncture after 12 h over-night fasting, without stasis in the sitting position. Whole-blood samples will be used for hematological evaluations. Most part of blood will be drawn into EDTA-containing tubes (1 mg/ml) and plasma will be isolated by centrifugation at 1000 xg, for 10 min and divided into aliquots of 250 μl for immediate analysis or for storage at -80 °C. Blood also will be used for obtaining isolated blood mononuclear cells (BMCs) for other additional analyses. Aliquots containing both, plasma or BMCs, will be preserved at -80º C until analyses.

Blood analyses will be as follows:

1. Biochemistry evaluations: fasting blood lipid levels (including high-density lipoprotein-cholesterol (HDL), low-density lipoprotein-cholesterol (LDL), direct LDL-cholesterol, very low density-cholesterol (VLDL) and triglycerides (TG), plasma glucose, high-sensitive C-reactive protein, LPa, cortisol, fibrinogen and homocysteine levels will be determined in plasma using an automatic analyzer. Patients showing fasting blood glucose > 126 mg/dL, using of antidiabetic medication or with a prior diagnosis of diabetes will be determined as Type 2 diabetes mellitus in accordance with the American Diabetes Association diagnostic criteria. Hypercholesterolemia will be defined as total serum cholesterol levels >200 mg/dL or use of lipid-lowering agents, according to the National Cholesterol Education Program Adult Treatment Panel III guidelines.
2. Hematological study: haemogram and blood cell profile in whole blood samples.
3. Circulating pro-inflammatory markers: circulating levels of multiple inflammatory cytokines including IL-1β and IL-18 will be analyzed by a commercial multiplex kit (Cytokine Panel 1B 25plex, Thermo Fisher Scientific). In addition, protein levels of active caspase-1 and gene expression of Nlrp3 (CIAS1) and caspase-1 will be determined in isolated PBMCs by Western-Blotting and RT-PCR, respectively, to evaluate inflammasome activity.
4. Autophagy markers: MAP-LC3, ATG12, p62, TFEB, Beclin-1 and B and D cathepsines levels will be determined by Western-Blotting in isolated PBMC protein isolates. Beclin-1, y Maplc3 gene expressions will be determined by RT-PCR in isolated PBMCs using beta-actin as housekeeper gene.
5. Oxidative stress markers and antioxidant capacity: damage to lipids will be analyzed through the determination in urine of 15-F2 isoprostanes, damage to proteins by determination of carbonyl proteins in plasma68 and damage to DNA through the determination in urine of 8-hydroxyguanosine (8OHdG). In addition, the determination of the in situ redox state will be performed in the subjects at the clinic by using a blood drop from a finger. It will be carried out through the Redoxsys system (Aytu BioScience, Inc., Englewood, USA), which also measures the antioxidant capacity of the sample. This is a novel system that measures with a reliability before not available the total redox charge in biological samples as well as the antioxidant capacity of them.
6. Metabolomic study: to carry out this analyses, the metabolites of the different samples are extracted first. Then the molecules present in the methanolic extract are separated by chromatography. The eluate is monitored in an ESI-Q-TOF-MS / MS system by electrospray98. The analysis of results will be carried out in collaboration with Dr. Reinald Pamplona, from the University of Lleida, with whom we have been collaborating on this issue for years and with whom we share a line of research and publications on metabolomics.

F) Periodontal microbiota study. Subgingival plaque samples will be collected from the three sites with the highest PPDs by putting on the periodontal pocket the tip of a filter paper during 30 s after isolating the zone.

Subgingival plaque samples collected in dry papers will be analyzed by PCR to evaluate the presence of known peridontopathogens: Phorphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Aggregatibacter actinomycetemcomitans, Prevotella intermedia, Fusobacterium nucleatum. The microbiota studies will be carried out using 16S rDNA mass sequencing techniques. Sequencing and bioinformatic analysis will be performed by the Integrated Microbiome Resource, from the University of Dalhousie, in Canada.

G) Determinations in urine.

Fasting urine will be collected and the following determinations will be performed:

1. Oxidative damage markers: 8-hydroxy-2-deoxyguanosine and total F2-isoprostanes will be measured in urine by a competitive enzyme immunoassay. Results will be normalized to urinary creatinine.
2. Oleuropein metabolites concentration: they will be quantified by LC-ESI-MS/MS as in previous studies.

H) Successful Aging Index calculus Successful aging index (SAI), with potential scores ranging from 0 to 10, will be employed to evaluate aging for study participants. The full index encompasses education, financial status, physical activity, BMI, GDS score, participation in social activities with friends, with family, yearly excursions, CVD risk factors score and Mediterranean diet adherence level to develop the index. A cumulative variable (range 0-4) indicating the overall burden of classical cardiovascular disease risk factors (i.e., obesity and history of hypertension, diabetes and hypercholesterolemia) will be developed (participants having none of the aforementioned risk factors will receive score 0, having one factor score 1, etc.).

I) Intervention success criteria To assess the success of the intervention with oleuropein, the reduction of 1 mm or more in probing depth (PD) will be taken as the main variable. In addition, and as secondary success criteria, a reduction of 1 mm or more in the attachment level will be taken, as well as a reduction of more than 20% in gingival bleeding on probing.

J) Statistic analysis A descriptive analysis of the main variables studied will be carried out. For normal quantitative variables, the mean and standard deviation will be calculated, or the median and percentiles in the case of non-normality. Qualitative variables will be expressed using absolute and relative frequencies. The normality of the variables will be checked with the Kolmogorov-Smirnov test in order to determine the need to carry out transformations (logarithmic and others) before carrying out the comparison studies. To study the effect of treatment on the different variables in the same group, the Student's t-test for related samples will be used. To carry out comparative analyzes at the same experimental time between both experimental groups, the Student's t-test for independent samples will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periodontitis, defined as interdental attachment loss in ≥2 non-adjacent teeth or lingual or buccal attachment loss ≥3 mm in ≥2 teeth.

Exclusion Criteria:

* Patients taking antimicrobial drugs in the previous 6 months or anti-inflammatory drugs during the previous 2 months,
* Patients taking regular vitamin supplementation,
* Patients receiving treatment for any periodontal condition,
* Patients with any autoimmune disease,
* Patients with any disease affecting oral mucosa,
* Patients with any systemic disease affecting bone metabolism,
* Patients with aggressive disease,
* Patients with physical or mental disability or unable to provide informed consent,
* Patients unable to swallow capsules,
* Patients at risk of complications from periodontal therapy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Probing depth | 120 days
  Change of 2 mm or more

SECONDARY OUTCOMES:
Attachment level | 120 days
  Change of 2 mm or more
Gum bleeding | 120 days
  Change of 20% or more

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Luis Quiles Morales, Granada, Spain

IPD SHARING:
Plan to Share IPD: No